CLINICAL TRIAL: NCT05950854
Title: 3D Joint Space Evaluation in Knee Osteoarthritis: The Importance of Weight-bearing and Flexion
Acronym: 3DJSW-MRI
Status: Recruiting | Type: Observational
Sponsor: Mylène Jansen (Other)
Collaborators: University of Twente (Other)
Responsible Party: Sponsor-Investigator, Mylène Jansen, Assistant Professor, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: 23-040
Record Dates: First submitted 2023-07-06; First posted 2023-07-18 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Weight-bearing MRI — Four MRI scans with 0.25T scanner: weight-bearing and non-weight-bearing with flexed and extended knee

SUMMARY:
Rationale: Osteoarthritis (OA) is mainly characterized by cartilage degeneration. In knee OA, measuring the distance between the tibia and femur, known as the joint space width (JSW), is an often-used method to quantify the progression of the disease or the effectiveness of treatments, because it is an indirect measure of cartilage degeneration. However, JSW is often measured while the patient is standing (weight-bearing) with slightly flexed knees, with a flexion angle of around 7-10 degrees, while direct cartilage thickness measurements are usually performed while the patient is lying down (non-weight-bearing) with an extended leg [1]. Because of this difference in positioning, it is difficult to compare different JSW and cartilage thickness measures, as it is not clear what happens with the JSW distribution in the joint when a patient changes position between weight-bearing/non-weight-bearing and flexion/extension. In this study, we aim to identify the changes that occur in the knee of OA patients under the influence of weight-bearing and/or flexion, to enable comparing joint space measures from different positions. In this research we want to use MRI as a three-dimensional imaging technique because there is no radiation involved..

Objective: To evaluate how the 3D knee joint space distribution in knee OA patients changes under the influence of weight-bearing (upright) and flexion MRI scanning.

Study design: Explorative cross-sectional study. Study population: 21 patients with symptomatic knee osteoarthritis (Kellgren-Lawrence grade 2 or 3) are included from the orthopaedics department of Medisch Spectrum Twente in Enschede.

Main study parameters/endpoints: The primary study parameter is the change in medial joint space width between the different positions (weight-bearing/non-weight-bearing and flexion/extension).

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic knee osteoarthritis in at least one knee
* > 18 years old
* Kellgren-Lawrence grade (severity) 2 or 3
* Good knowledge of the Dutch language
* Signed informed consent

Exclusion Criteria:

* Previous surgery in (both) symptomatic knee(s)
* Inability to stand for 15 minutes, without assistance
* Unable to fit knee in the MRI coil (knee width > ~15 cm)
* Not eligible for MRI, in response to the MRI safety checklist

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic and radiographic (Kellgren-Lawrence grade 2-3) knee osteoarthritis eligible for MRI scanning
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Medial joint space width | 1 hour
  Medial joint space width in four scan positions

SECONDARY OUTCOMES:
Lateral joint space width | 1 hour
  Lateral joint space width in four scan positions

CONTACTS AND LOCATIONS:
Overall Officials: Wyger Brink, PhD, Principal Investigator — University of Twente; Simon Mastbergen, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University of Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided